CLINICAL TRIAL: NCT02209090
Title: Randomised Clinical Trial: Modified Intrapartum Maternal Sims Position-related Efficiency in the Correction of Persistent Foetal Occipito-posterior Position
Brief Title: Modified Intrapartum Sims Position-related Efficiency in Correction of Persistent Foetal OP Positions
Acronym: MSIMSFPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AMI)182/2012
Record Dates: First submitted 2014-07-02; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Persistent Occiput Posterior Position During Labor
Keywords: occiput-posterior; occipitoposterior; labour

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- maternal modified sims position (Experimental): Women in this group will adopt the modified Sims position, lying on the side of the foetal back.
  This position is maintained for the greater part of labour, at least 40 minutes, every hour. The mother can use other positions during resting time of no more than 20 minutes each hour, but never use a lateral position against the side of the foetal back.
  Interventions: Procedure: maternal modified sims position
- maternal free positions (Sham Comparator): Women can adopt the position they wish and which is most comfortable, except for lateral positions which can only be used for a maximum of 20 minutes each hour to avoid confounding factors.
  Interventions: Procedure: maternal free positions

INTERVENTIONS:
Procedure: maternal modified sims position — Maternal Modified Sims position during at least 40 minutes for each 60 minutes
  Arms: maternal modified sims position
Procedure: maternal free positions — At least 40 minutes each hour during labour
  Arms: maternal free positions

SUMMARY:
Aim: To evaluate the efficiency of the modified Sims position versus maternal free positions in the rotation of persistent foetal occipito-posterior position intrapartum in pregnant women with epidural anaesthesia.

Design: An open, randomised, controlled and parallel clinical trial will be conducted at the Delivery Room of the Area Materno-Infantil, Hospital Universitari Vall d'Hebron, Barcelona, Spain.

Method: Fifty-six pregnant women with persistent foetal occipito-posterior position will be selected. Each woman will be assigned to a control or experimental group via an opaque envelope at a 1:1 ratio.

The control group will deliver in free intrapartum positions, and the experimental group in a modified Sims position. Correction of foetal position is the key study variable, and delivery type the secondary variable. Statistical analyses will be made with the SPSS v.20 program.

DETAILED DESCRIPTION:
Aim: To evaluate the efficiency of the modified Sims position versus maternal free positions in the rotation of persistent foetal occipito-posterior position intrapartum in pregnant women with epidural anaesthesia.

Background: There is a theoretical basis for the possible effects of maternal positions on foetal positions. Despite all the studies published in recent years, conclusive trials providing significant scientific evidence are lacking.

Design: An open, randomised, controlled and parallel clinical trial will be conducted at the Delivery Room of the Area Materno-Infantil, Hospital Universitari Vall d'Hebron, Barcelona, Spain.

Method: Fifty-six pregnant women with persistent foetal occipito-posterior position will be selected. Each woman will be assigned to a control or experimental group via an opaque envelope at a 1:1 ratio.

The control group will deliver in free intrapartum positions, and the experimental group in a modified Sims position. Correction of foetal position is the key study variable, and delivery type the secondary variable. Statistical analyses will be made with the SPSS v.20 program.

Discussion: If the modified maternal Sims position proved to correct persistent foetal occipito-posterior positions and being a non-invasive, low-cost, non-prejudicial method for both mother and foetus, maternal and foetal morbidity problem would be reduced

ELIGIBILITY:
Inclusion Criteria:

* adult pregnant women (>18 years of age)
* persistent posterior foetal position diagnosed during labour through two vaginal examinations two hours apart.
* at-term gestations (37 to 42 weeks)
* women in labour with epidural anaesthesia

Exclusion Criteria:

* multiple gestations
* previous severe foetal malformation diagnosed
* macrosomic foetus diagnosed by ultrasound in the 3rd trimester (> percentile 95), or IUGR (< percentile 10)
* women with contraindicated vaginal delivery owing to previous vaginal surgeries
* women with severe heart diseases
* diabetic pregnant women (types I, II and gestational)
* hypertension problems during labour
* myopathies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Rotation | During labour
  the foetal head's capacity to rotate 145º clockwise until the minor fontanelle is situated under the pubic bone, expressed as yes or no, depending on whether there is rotation or not.

SECONDARY OUTCOMES:
rotating to OA | During labour
  length of time taken by the foetal head to reach OA expressed in minutes from the start of the intervention
Delivery mode | The first two hours after delivery
  eutocic: vaginal delivery, foetal head expulsion in vertex position, spontaneous

OTHER OUTCOMES:
uterine dynamics | During labour
  assessed by frequency and intensity according to Monteviedo unit calculation
first stage in minutes | During labour
  timed in minutes, from 3cm with cervix shortened until complete diltation.
second stage in minutes | The first two hours after delivery
  timed from complete dilation to foetal head expulsion
epidural anaesthesia | During labour
  doses of epidural anaesthesia required, concentration and ml.
episiotomy | The first two hours after delivery
  whether performed or not to gain a major opening from the soft parts of the birth canal.
tear | The first two hours after delivery
  trauma occurring spontaneously by the foetal head passing through the vaginal cavity and/or perineum:
reason to end labour earlier | The first two hours after delivery
  cause that occurs on ending labour before it concludes spontaneously. Reasons may be foetal: risk of loss of foetal wellbeing, or maternal: pelvic foetal disproportion or stopped labour
maternal comfort during labour | The first two hours after delivery
  MACKEY SATISFACTION CHILDBIRTH RATING SCALE validated in Spanish

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bueno, PhDcandidate, Principal Investigator — HUValldebronRI
Locations (1):
- Area Materno Infantil of the Hospital Univeristario Vall d'Hebron (AMI HUVH),, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Bueno-Lopez V, Fuentelsaz-Gallego C, Casellas-Caro M, Falgueras-Serrano AM, Crespo-Berros S, Silvano-Cocinero AM, Alcaine-Guisado C, Zamoro Fuentes M, Carreras E, Terre-Rull C. Efficiency of the modified Sims maternal position in the rotation of persistent occiput posterior position during labor: A randomized clinical trial. Birth. 2018 Dec;45(4):385-392. doi: 10.1111/birt.12347. Epub 2018 Mar 14. PMID 29537658